CLINICAL TRIAL: NCT04851535
Title: A Phase II Study To Evaluate The Efficacy And Safety of Jaktinib Hydrochloride Tablets In Patients With Myelofibrosis Who Were Relapsed or Refractory of Ruxolitinib Treatment
Brief Title: Study of Jaktinib In Patients With Myelofibrosis Who Were Relapsed or Refractory of Ruxolitinib Treatment.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZGJAK017
Record Dates: First submitted 2021-04-08; First posted 2021-04-20 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Jaktinib 100mg Bid (Experimental): Jaktinib twice daily for 6 consecutive 28-day cycles, orally, empty stomach
  Interventions: Drug: Jaktinib Hydrochloride Tablets

INTERVENTIONS:
Drug: Jaktinib Hydrochloride Tablets — Jaktinib 100mg Bid

SUMMARY:
This was a phase 2, single-arm, open-label, non-randomised, multicentre, study to evaluate the efficacy and safety of Jaktinib in patients with myelofibrosis who were relapsed or refractory of ruxolitinib treatment.

DETAILED DESCRIPTION:
All subjects will receive a minimum of 6 treatment cycles or 24 weeks (a 28-day treatment cycle is defined as one treatment cycle).

ELIGIBILITY:
Inclusion Criteria:

* Subjects voluntarily sign the informed consent form (ICF);
* Age ≥ 18 years, either male or female;
* Subjects diagnosed with a PMF according to World Health Organization (WHO) criteria (2016 Edition), or patients diagnosed with a Post-PV-MF or Post-EF-MF according to International Working Group for Myeloproliferative Neoplasms Research and Treatment (2007 IWG-MRT) criteria;
* Subjects with intermediate-2 or high-risk myelofibrosis, or Intermediate-1 myelofibrosis with symptoms according to the Dynamic International Prognostic System (DIPSS) scoring system;
* Subjects are relapsed/refractory to Ruxolitinib:

  1. Relapsed defined as Ruxolitinib treatment for ≥ 3 months, following an initial response, regrowth to < 10% spleen volume reduction (SVR) by MRI or < 30% decrease in spleen size by palpation from baseline;
  2. Refractory defined as Ruxolitinib treatment for ≥ 3 months observed inadequate efficacy response: < 10%volume SVR by MRI or < 30% decrease in spleen size by palpation from baseline.
* Subject has a measurable splenomegaly: spleen volume of ≥ 450 cm3 by MRI/CT and ≥ 5 cm below left costal margin by palpation spleen measuring;
* Expected life expectancy is greater than 24 weeks;
* Eastern Cooperative Oncology Group (ECOG) performance Score 0-2;
* Laboratory examination within 7 days before the randomization, fulfilling the following criteria:

Neutrophil count ≥ 0.75 x 109/L, platelet count ≥ 75 x 109/L; Peripheral blood blasts ≤ 10%; ALT and AST≤ 3 ULN, DBIL ≤ 2.0 ULN; Serum creatinine ≤ 2.0 ULN.

Exclusion Criteria:

* Subjects who have been previously exposed to Janus kinase (JAK) inhibitors other than Ruxolitinib for a total of> 2 weeks;
* Subjects who have taken Ruxolitinib or other JAK inhibitor within 1 week prior to screening;
* Subjects with any significant clinical and laboratory abnormalities which may affect the safety evaluation, such as uncontrolled diabetes, uncontrolled hypertension after taking two or more hypotensive drugs or peripheral neuropathy;
* Subjects with congestive heart failure (NCI-CTCAE V5.0) Class II or above, uncontrolled or unstable angina or myocardial infarction, cerebrovascular accident, or pulmonary embolism within 6 months prior to screening;
* Subjects who have a history of chronic or recurrent respiratory diseases, such as: chronic obstructive pulmonary disease, recurrent lung infections, etc., or have a history of lung infections within 3 months before screening, or currently have upper respiratory tract infections that have not recovered;
* Subjects who have not fully recovered from surgical operation within 4 weeks prior to screening;
* Subjects suffering from arrhythmia and requiring treatment, or QTcB > 480ms at screening;
* Subjects with clinical symptoms of active bacterial, viral, parasitic or fungal infections requiring treatment at screening;
* Subjects who had undergone splenectomy, or received radiotherapy to the spleen within 6 months before screening;
* Subjects with known human immunodeficiency virus (HIV), known active infectious Hepatitis B (HepB), and/or known active infectious Hepatitis C (HepC);
* Female subjects who are pregnant, currently breastfeeding, planning to become pregnant;
* Subjects who had experienced malignant tumors (except for adequately treated local basal cell or squamous cell carcinoma of the skin and cervical carcinoma in situ that have been cured) or in combination with other serious diseases within the past 5 years;
* Subjects who have participated in another clinical trial of a new drug or medical instrument within 1 month before screening.
* Subjects who have any other conditions that are not specified in the protocol but the investigator believes that they are not suitable for inclusion in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Spleen Volume Response rate (SVRR) at Week 24 | at Week 24
  The proportion of subjects with spleen volume reduction from baseline ≥ 35% measured by MRI or CT.

SECONDARY OUTCOMES:
Clinical Objective Response Rate (complete remission (CR) + partial remission (PR)) | Baseline, up to Year 2
  International Working Group for Myeloproliferative Neoplasms Research and Treatment (IWG-MRT) response criteria.
Spleen Response | up to Year 2
  Best response rate: the proportion of subjects with at least one spleen volume reduction ≥ 35% against the baseline; Time to response: the length of time from the date of first dose to the date on which the first spleen volume reduction ≥ 35% against the baseline; Duration of maintenance of at least 35% Reduction in Spleen Volume (DoMSR): the length of time from the date of the first spleen volume reduction ≥ 35% against the baseline to the date of the spleen volume reduction is less than 35% against the baseline due to spleen volume increase.
Anemia Response | up to Year 2
  Proportion of transfusion dependent patients（Transfusion dependent patients：received RBC transfusion ≥ 12 U within 12 weeks before receiving the investigational drug） at baseline turned to non-transfusion dependent patients (non-transfusion dependent patients: no transfusion for at least 12 consecutive weeks and Hgb ≥ 85 g/L); Proportion of hemoglobin (Hgb) elevation ≥ 20 g/L in non-transfusion dependent patients (Hgb ≤ 100 g/L) at baseline; Decline in red blood cell (RBC) transfusion dependence: Number of RBC transfusions decreases by 50%.
Response rate of MF-related symptoms | Baseline, up to Year 2
  Proportion of patients with Myeloproliferative neoplasm symptom assessment form (MPN-SAF) TSS decreasing from baseline by ≥ 50%; The change in MPN-SAF TSS from baseline.
Progression free survival (PFS) | From the date of first dose to the earliest date of either increase in spleen volume ≥ 25% from on-study nadir or death, up to Year 2
  The length of time from the date of first dose to the date of any of the following events: 1) ≥ 25% increase in spleen volume over nadir since the treatment; 2) death from any cause.
Leukemia free survival (LFS) | From the date of first dose to the earliest date of either leukemia or death, up to Year 2
  The length of time from the date of first dose to the date of any of the following events: 1) the first bone marrow blast count ≥ 20%; 2) the first peripheral blast count ≥ 20% ; 3) death from any cause.
Overall survival (OS) | From the date of first dose to the date of death, up to Year 2
  The length of time from the date of first dose to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Jin, PhD, Principal Investigator — Zhejiang University
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China